CLINICAL TRIAL: NCT07223047
Title: A Phase 1/2a, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of BMS-986523 As Monotherapy and in Combination With Anti-Cancer Agents in Participants With Advanced Solid Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of BMS-986523 Alone and in Combination With Anti-Cancer Agents in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA256-0001; 2025-523547-35 (Other: EU CTR)
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Malignancies; Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma (PDAC); Pancreatic Cancer; Lung Cancer; Kirsten rat sarcoma viral oncogene homolog (KRAS)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental)
  Interventions: Drug: BMS-986523
- Arm B (Experimental)
  Interventions: Drug: BMS-986523
- Arm C (Experimental)
  Interventions: Drug: BMS-986523
- Arm D (Experimental)
  Interventions: Drug: BMS-986523; Drug: Pembrolizumab
- Arm E (Experimental)
  Interventions: Drug: BMS-986523; Drug: Cetuximab
- Arm F (Experimental)
  Interventions: Drug: BMS-986523; Drug: Gemcitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: BMS-986523 — Specified dose on specified days
Drug: Gemcitabine — Specified dose on specified days
  Arms: Arm F
Drug: Nab-Paclitaxel — Specified dose on specified days
  Arms: Arm F
Drug: Cetuximab — Specified dose on specified days
  Arms: Arm E
Drug: Pembrolizumab — Specified dose on specified days
  Arms: Arm D

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of BMS-986523 alone and in combination with anti-cancer agents in participants with advanced solid malignancies

ELIGIBILITY:
Inclusion Criteria

* Participants must have a histologically confirmed diagnosis of a locally advanced and unresectable or metastatic solid tumor malignancy with a known Kirsten rat sarcoma viral oncogene homolog (KRAS) alteration (mutation or amplification).
* Participants must, for Arm D, have a PD-L1 expression (≥50%).
* Participants must have previously received, be ineligible for, or decline (after having been provided adequate information to make an informed decision) the protocol defined standard of care (SoC) treatments.

Exclusion Criteria

* Participants must not have untreated central nervous system (CNS) metastases.
* Participants must not have concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to treatment.
* Participants must not have a history of, or any evidence of, interstitial lung disease or active, non-infectious pneumonitis. A history of radiation pneumonitis in the radiation field is permitted.
* Participants must not have a history of prior severe cutaneous adverse reactions (SCARs), including Stevens-Johnson Syndrome (SJS) and toxic epidermal necrolysis (TEN).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-10-13 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 3 years
Number of participants with serious adverse events (SAEs) | Up to 3 years
Number of participants with AEs meeting protocol-defined dose limiting toxicity (DLT) criteria | Up to 3 years
Number of participants with AEs leading to discontinuation | Up to 3 years
Number of deaths | Up to 3 years

SECONDARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the investigator. | Up to 3 years
Duration of response (DOR) per RECIST v1.1 as assessed by the investigator. | Up to 3 years
Maximum observed plasma concentration (Cmax) | Up to 3 years
Time of maximum observed plasma concentration (Tmax) | Up to 3 years
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (4):
  - Local Institution - 0009, Baltimore, Maryland
  - NEXT Oncology, San Antonio, Texas
  - Local Institution - 0007, Salt Lake City, Utah
  - Local Institution - 0011, Fairfax, Virginia
- Canada (2):
  - Local Institution - 0002, Vancouver, British Columbia
  - Local Institution - 0010, Toronto, Ontario
- Spain (2):
  - Local Institution - 0006, Badalona, Barcelona [Barcelona]
  - Local Institution - 0008, Hortaleza, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07223047.html